CLINICAL TRIAL: NCT06923462
Title: VoiceLove: An App-Based COMMunication Tool Designed to Address DeliriUm and Improve Family ENgagement and PatIent/Family SatisfaCtion in CriticAlly Ill PaTiEnts (COMMUNICATE)
Acronym: COMMUNICATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wes Ely, Co-Director, CIBS Center, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 242209
Record Dates: First submitted 2025-03-06; First posted 2025-04-11 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Intensive Care Medicine
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care recipients (No Intervention): Participants in this arm will be randomized to usual care, or no VoiceLove utilization while in the ICU.
- VoiceLove recipients (Experimental): Participants in this arm will be randomized to utilize VoiceLove while in the ICU.
  Interventions: Other: Communication Application

INTERVENTIONS:
Other: Communication Application — Participants will receive the VoiceLove intervention versus the standard care which does not utilize VoiceLove.
  Arms: VoiceLove recipients

SUMMARY:
VoiceLove is a phone application allowing family and patients to share information in a secure platform. This project will compare the VoiceLove app to usual care to learn about whether VoiceLove improves patient-family communication, family engagement, and ICU delirium.

DETAILED DESCRIPTION:
VoiceLove is a novel, HIPAA compliant mobile phone application that enables families and patients to securely exchange and archive voice messages in real-time. For patients who are intubated or otherwise unable to communicate, VoiceLove allows family members to deliver real-time voice messages when they are away from the bedside without relying on the clinical team to coordinate calls. The investigator group has recently completed formative usability testing of the VoiceLove application with a variety of ICU stakeholders including family members, bedside ICU nurses, and ICU physicians to refine and optimize the app for clinical use in the ICU. During usability testing, stakeholders overall viewed the app favorably and expressed interest in tools to enhance communication in the ICU. As compared to traditional methods of communication, stakeholders identified the ability to customize messaging by unique family groups and to archive and replay messages as strengths. While promising as a tool to improve family engagement in the ICU, it has yet to undergo evaluation in the ICU to assess feasibility and acceptability of use.

The goal in this prospective, mixed method randomized control trial (RCT) is to compare VoiceLove implementation to usual care to investigate the effect of VoiceLove on optimizing patient-family communication, family engagement, and ICU delirium prevalence.

ELIGIBILITY:
Inclusion Criteria

Only patients who meet inclusion criteria, have no exclusion criteria, and consent for participation will advance to the Interventional Trial phase (i.e., the randomization phase) of the study. Patients will be eligible for inclusion in the Pre-Randomization Phase of the study (i.e., presented for study consent) if they are:

1. Adult patient ≥18 years old
2. Admitted to medical or coronary ICU
3. Intubated on mechanical ventilation with expected intubation of > 24 hours

Exclusion Criteria

Patients will be excluded (i.e., not consented) for any of the following reasons:

1. Inability to obtain informed consent

   * Attending physician refusal
   * Patient and/or surrogate refusal
   * Patient unable to consent and no surrogate available
2. Acute or chronic neurologic deficit precluding CAM-ICU assessments
3. Inability to understand English
4. Current enrollment in a study that does not allow co-enrollment
5. Prisoners
6. Expected death or comfort measures within 24 hours of enrollment or lack of commitment to intervention by family or the medical team (e.g., likely to withdraw life support measures within 24 hours of enrollment).
7. Bilateral Deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Assess engagement among patients during acute hospitalization | Up to 14 days
  Within the intervention group and control groups, engagement will be assessed through survey administered at ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: E Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plans for sharing data are being developed.